CLINICAL TRIAL: NCT03052647
Title: Comparison of Adhesive Latch Device to Subcuticular Skin Closure at the Time of Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rubino Ob-Gyn Group (Other)
Responsible Party: Principal Investigator, Robert J. Rubino, MD, FACOG, Principal investigator , Assistant Clinical Professor, Rubino Ob-Gyn Group
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Rubinoobgyn
Record Dates: First submitted 2017-02-03; First posted 2017-02-14 (Actual); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Wound
Keywords: dermaclip; subcuticular; cesarean section; staples; adhesive latch; rousseau
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: A control group of subcuticular closure and the experimental group is skin closure withthe adhesive latch device ("dermaclip")
Who Masked: Participant, Investigator
Masking Description: computer randomized list of closure type opened from a sealed envelope on the day of surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Subcuticular arm (Active Comparator): closure technique that the Adhesive Latch arem (dermaclip) arm is being compared to
  Interventions: Device: Subcuticular suture
- Adhesive Latch Arm (Demaclip arm) (Active Comparator): This is the arm which the adhesive latch system is used and it is being compared to the arm of subcuticular
  Interventions: Device: Dermaclip

INTERVENTIONS:
Device: Dermaclip — Dermaclip is an adhesive latch device used for skin closure
  Other Names: adhesive latch device, dermaclip
  Arms: Adhesive Latch Arm (Demaclip arm)
Device: Subcuticular suture — subcuticular suture will be used as the device to close the skin in this arm
  Other Names: sucuticular
  Arms: Subcuticular arm

SUMMARY:
The objective of this study was to compare the an adhesive latch device (" Dermaclip") to subcuticular skin closure at the time of cesarean section. Currently, no studies exist comparing these two closure techniques. The hypothesis is dermaclip closure is faster than subcuticular closure. The null hypothesis is there is no difference in closure times. There is a study (see reference at bottom) that compares staples closure to subcuticular closure, but none comparing subcuticular to dermaclip closure. Dermaclip device is easily deployed and is expected to be as fast as staples closure compared to subcuticular as noted in the prior study referenced below.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18
2. Elective cesarean section
3. Term pregnancy

Exclusion Criteria:

1. Fever >101F in the past 14 days
2. Antibiotics in the past 14 days
3. Suspected ongoing infection
4. Poorly controlled gestational diabetes
5. Allergic to adhesive

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-11-30 (Estimated); Study Completion 2018-03-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of adhesive latch device to subcuticular skin closure at the time of cesarean section | 18 months
  The time for skin closure between subcuticular and demaclip techniques will compared during cesarean section

SECONDARY OUTCOMES:
Pain Scores | 18 months
  - pain scores using the visual analog pain scale (VAPS) system
Wound Infections as measured in centimeters of erythema | 18 months
  - wound infections will measured in centimeters of redness/erythema around the infected area
Wound separation as measured in centimeters | 18 months
  - wound separation will be recorded centimeters
Patient Satisfaction scores | 18 months
  - patient satisfaction
Total surgery time | 18 months
  - total surgery time
Age | 18 months
  - age (years)
BMI | 18 months
  BMI of participants bmi (in kg/m2, weight in kg, height, in meters)
Ethnicity | 18 months
  Ethnic origin
Race | 18 months
  Race of participants

CONTACTS AND LOCATIONS:
Locations (1):
- Rubino OBGYN Group, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No